CLINICAL TRIAL: NCT05598281
Title: An Open-label, Drug-drug Interaction Study to Evaluate the Effect of AMG 510 on the Pharmacokinetics of Digoxin, a P-glycoprotein Substrate, in Healthy Subjects
Brief Title: Study to Evaluate the Effect of AMG 510 on the Pharmacokinetics (PK) of Digoxin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20190315
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Healthy Participants
Keywords: AMG 510; Healthy Participants; Digoxin
MeSH Terms: interventions — sotorasib; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AMG 510 + Digoxin (Experimental): Participants will receive digoxin on Day 1 and both AMG 510 + digoxin on Day 7.
  Interventions: Drug: AMG 510; Drug: Digoxin

INTERVENTIONS:
Drug: AMG 510 — Oral tablet
  Other Names: Sotorasib
Drug: Digoxin — Oral tablet

SUMMARY:
The primary objective of the study is to evaluate the PK of digoxin administered alone and in combination with AMG 510 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects or female subjects, between 18 and 60 years of age (inclusive), at the time of Screening.
* Body mass index, between 18 and 30 kg/m2 (inclusive), at the time of Screening.
* Females of nonchildbearing potential.

Exclusion Criteria:

* Inability to swallow oral medication or history of malabsorption syndrome.
* History of hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee) and in consultation with the Sponsor.
* Poor peripheral venous access.
* History or evidence, at Screening or Check in, of clinically significant disorder, condition, or disease not otherwise excluded that, in the opinion of the Investigator (or designee), would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2019-11-19 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of Digoxin Administered Alone | Day 1
Area Under the Plasma Concentration-time Curve (AUC) from Time Zero to Time of Last Quantifiable Concentration (AUClast) of Digoxin Administered Alone | Day 1
AUC from Time Zero to Infinity (AUCinf) of Digoxin Administered Alone | Day 1
Maximum Plasma Concentration (Cmax) of Digoxin Administered in Combination with AMG 510 | Day 7
AUClast of Digoxin Administered in Combination with AMG 510 | Day 7
AUCinf of Digoxin Administered in Combination with AMG 510 | Day 7

SECONDARY OUTCOMES:
Number of Participants with an Adverse Event (AE) | Day 1 to Day 13
  Any clinically significant changes in clinical laboratory tests, 12-lead electrocardiograms and vital signs will be recorded as AEs.
Cmax of AMG 510 Administered in Combination with Digoxin | Day 7
AUClast of AMG 510 Administered in Combination with Digoxin | Day 7
AUCinf of AMG 510 Administered in Combination with Digoxin | Day 7

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Covance Clinical Research Unit, Inc, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com